CLINICAL TRIAL: NCT03084250
Title: A Prospective, Randomized, Open-label Study of the Investigation of Peginterferon Alfa-2a on Optimal in Chronic Hepatitis B Patients Who Have a High Risk of HCC
Brief Title: The Investigation of Peginterferon Alfa-2a on Optimal in Chronic Hepatitis B Patients Who Have a High Risk of HCC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Nanhui Nanhua Hospital (Other)
Responsible Party: Principal Investigator, Chenbo Hu, Dr.Chenbo Hu, Shanghai Nanhui Nanhua Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: High risk of HCC
Record Dates: First submitted 2017-03-14; First posted 2017-03-20 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — peginterferon alfa-2a; adefovir; entecavir; Tenofovir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination (Experimental): The subjects will be treated by nucleotide analogue (NA) combination with peginterferon alfa-2a
  Interventions: Drug: Peginterferon Alfa-2A
- nucleotide analogue (Active Comparator): The subjects will be treated by nucleotide analogue (NA) only
  Interventions: Drug: Adefovir, entecavir,tenofovir, either of them

INTERVENTIONS:
Drug: Peginterferon Alfa-2A — 180μg/week, 48 weeks; 135μg/week,48weeks
  Other Names: Pegasys
  Arms: Combination
Drug: Adefovir, entecavir,tenofovir, either of them — Adefovir, entecavir,tenofovir, either of them is ok
  Arms: nucleotide analogue

SUMMARY:
The CHB subjects who are cirrhosis, will be randomized to two groups.

The subjects who go into group A will be treated by nucleotide analogue (NA) combination with peginterferon alfa-2a,180μg/week for 48 weeks.

The subjects who go into group B will be treated by nucleotide analogue (NA) only for 48 weeks.

DETAILED DESCRIPTION:
This study is a prospective, randomized, open-label study.

The CHB subjects who are cirrhosis will be randomized to two groups.

The subjects who go into group A will be treated by nucleotide analogue (NA) combination with peginterferon alfa-2a,180μg/week for 48 weeks.

The subjects who go into group B will be treated by nucleotide analogue (NA) only for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients with age ≥18 and ≤65 years;
2. There should be evidences that HBsAg has been positive for more than 6 months with HBsAb and HBeAb negative; HBV-related cirrhosis
3. Women without ongoing pregnancy or breast feeding and both women and men willing to take an effective contraceptive measure during the treatment;
4. Agree to participate in the study and sign the patient informed consent form.

Exclusion Criteria:

1. Treated by immunosuppressant,immunomodulator,Systemic cytotoxic drug,herbs or HBIg within 6 months prior to the first dose of treatment;
2. ALT≥10 X ULN or total bilirubin ≥2 X ULN;
3. Allergic history to interferon;
4. Co-infection with active hepatitis A, hepatitis C, hepatitis D and/or human immunodeficiency virus (HIV);
5. Child-Pugh scores >7;
6. History or other evidence of a medical condition associated with chronic liver disease other than viral hepatitis (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures, thalassemia);
7. Pregnant or breast-feeding Women;
8. Consuming alcohol in excess of 20g/day for women and 30g/day for men within 6 months prior to enrollment or drug taking history;
9. ANC(absolute neutrophil count)<1.5x 10^9/L or PLT(platelet count)<90x 10^9/L
10. Creatinine over upper limit of normal;
11. History of severe psychiatric disease, especially depression. Severe psychiatric disease is defined as major depression or psychosis that treated with antidepressant medication or a major tranquilizer at therapeutic doses respectively at any time prior to 3 months or any history of the following: a suicidal attempt hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease;
12. History of immunologically mediated disease, (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, scleroderma, rheumatoid arthritis etc.);
13. History of esophageal varices bleeding or other evidence of esophageal varices bleeding or other symptoms consistent with decompensated liver disease;
14. History of severe cardiac disease (e.g., New York Heart Association Functional Class III or IV, myocardial infarction within 6 months, ventricular tachyarrhythmias requiring ongoing treatment, unstable angina or other significant cardiovascular diseases);
15. Hemodialysis patients or patients with renal insufficiency;
16. History of a severe seizure disorder or current anticonvulsant use;
17. Major organ transplantation or other evidence of severe illness, malignancy, or any other conditions, which would make the patient, in the opinion of the investigator, unsuitable for the study;
18. History of thyroid disease poorly controlled on prescribed medications;
19. Evidence of severe retinopathy or clinically relevant ophthalmologic disorder;
20. History of other severe disease or evidence of other severe disease or any other illness or conditions that the investigator believe that patients are not suitable to join in the study;
21. Patients included in another trial or having been given investigational drugs within 12 weeks prior to screening;
22. AFP(alpha feto protein)>50ng/ml and/or evidence of hepatocellular carcinoma;
23. Patients treated with Telbivudine;
24. Other disease should exclusive considered by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-03-10 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of subjects who develop to hepatocellular carcinoma during 5 years | 5 years
  The number of subjects develop to hepatocellular carcinoma during 5 years will be measured

SECONDARY OUTCOMES:
Number of participants who achieve HBeAg loss and HBeAg seroconversion | year 1,2,3,4,5
  The number of subjects with HBeAg loss and HBeAg seroconversion at year 1 ,2,3,4 and 5 will be measured
Number of participants who achieve HBsAg loss and HBsAg seroconversion | year 1,2,3,4,5
  The number of subjects with HBsAg loss and HBsAg seroconversion at year 1, 2,3,4 and 5 will be measured
The factor such as HBsAg level related to the incidence of HCC development | year 1
  The HBsAg level at year 1 will be measured, to assess whether the quantitative HBsAg level related to the incidence of HCC development

CONTACTS AND LOCATIONS:
Overall Officials: Chenbo Hu, Principal Investigator — Nanhua Hospital
Locations (1):
- Nanhua Hospital, Shanghai, China